CLINICAL TRIAL: NCT07304596
Title: Evaluation of Responsiveness of Hindi Version of Oral Health Impact Profile for Periodontitis (OHIP-P-HIN)
Brief Title: Responsiveness of Hindi Version of Oral Health Impact Profile for Periodontitis (OHIP-P-HIN)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Navi Bansal Periodontics
Record Dates: First submitted 2025-12-02; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis; Oral Health Quality of Life (OHQoL) Was Assessed
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non Surgical Periodontal Therapy (Other): Full mouth Sub gingival instrumentation will be done
  Interventions: Procedure: Non Surgical Periodontal Therapy

INTERVENTIONS:
Procedure: Non Surgical Periodontal Therapy — Full mouth subgingival instrumentation will be done

SUMMARY:
The distribution- and anchor-based methods will be used to estimate the Minimal Important Difference (MID) of the OHIP-P-HIN. Two established distribution-based approaches, the standardized effect size (ES) and standardized response mean (SRM) will be calculated. The ES is calculated by dividing the mean change scores in the OHIP-P-HIN from baseline by the standard deviation of the baseline scores. And the SRM are computed as ratios of the mean change score divided by its standard deviation. The anchor-based approach will be applied by using the global transition scale as the anchor.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* patients able to understand and complete questionnaires independently
* confirmed diagnosis of periodontitis

Exclusion Criteria:

* Patients with systemic diseases such as acquired immunodeficiency syndrome or diabetes mellitus
* pregnancy
* required prophylactic antibiotic coverage prior to dental treatment,
* patients with bleeding disorders
* patients who had received non-surgical periodontal therapy within the preceding eight weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Minimal Important Difference (MID) | 6 weeks after completion of Non surgical Periodontal therapy
  The distribution- and anchor-based methods will be used to estimate the MID. Two established distribution-based approaches, the standardized effect size (ES) and standardized response mean (SRM) will be calculated. The anchor-based approach will be applied by using the global transition scale as the anchor.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS Rohtak, Rohtak, Haryana, India